CLINICAL TRIAL: NCT00394082
Title: A Phase II Trial of Weekly Administration of ABI-007 In Combination With Bevacizumab in Women With Metastatic Breast Cancer
Brief Title: ABI-007 In Combination With Bevacizumab in Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA043
Record Dates: First submitted 2006-10-30; First posted 2006-10-31 (Estimated); Results first posted 2013-05-22 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer, Abraxane, Bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; 130-nm albumin-bound paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABI-007 plus Bevacizumab (Experimental): ABI-007 is administered on days 1, 8 and 15 at 125 mg/m^2 and bevacizumab is administered on day 1 and 15 at 10 mg/kg of each 28 day cycle. Treatment continues until disease progression or intolerable toxicity. If a patient develops intolerable toxicity to only one of the drugs, the other drug may be continued as single agent therapy in the absence of progression, as long as the treating physician feels this is in the best interests of the patient.
  Interventions: Drug: ABI-007; Drug: Bevacizumab

INTERVENTIONS:
Drug: ABI-007 — 125 mg/m^2 of ABI-007 administered by intravenously (IV) over 30 minutes on days 1, 8 and 15 of each 28 day cycle.
  Other Names: Abraxane®; Nab-paclitaxel
Drug: Bevacizumab — Bevacizumab administered once every 2 weeks (10 mg/kg) by IV infusion after ABI-007 has been given. The first dose is one Day 1, cycle 1.
  Other Names: NSC 704865; RhuMAb VEGF; Recombinant Humanized Monoclonal Bevacizumab Antibody

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of weekly ABI-007 in combination with bevacizumab.

The evaluation of progression-free survival of weekly ABI-007 in combination with bevacizumab for patients with previously untreated advanced/metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the breast.
* Stage IV disease.
* Measurable disease (defined as the presence of at least one lesion that can be accurately measured in at least one dimension with longest diameter greater or = 1.0 cm with spiral computed tomography (CT) scan).
* Patients must not be a candidate for Herceptin therapy (i.e., patients with HER-2 positive disease (gene amplification by fluorescence in situ hybridization (FISH) or 3 + overexpression by ICH) and patients with unknown HER-2 status are ineligible unless the treating physicians has determined that Herceptin-based therapy would be inappropriate or not indicated).
* For subjects with prior anthracycline exposure, normal cardiac function including a baseline left ventricle ejection fraction >50% or above institution's lower limit of normal and a normal electrocardiogram (ECG) (as assessed by the investigator).
* At least 2 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation portal or there must be pathologic proof of progressive disease within the radiation portal.
* International Normalized Ratio (INR) < 1.5 and activated partial thromboplastin time within normal limits (APTT WNL).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Female > 18 years of age.
* Patients have the following blood counts at Baseline: absolute neutrophil count (ANC) greater or equal to 1.5 x 10^9 cells/L; platelets greater or equal 100 x 10^9 cells/L; hemoglobin (Hgb) greater or equal to 9g/dL.
* Patients have the following blood chemistry levels at Baseline: aspartate aminotransferase (AST or SGOT), alanine aminotransferase (ALT or SGPT) less than or equal 2.5x upper limit of normal (ULN) range (less than or equal 5x ULN if patient has known liver metastases); total bilirubin greater than or equal to ULN; creatinine greater or equal to 1.5mg/dL.
* if female of childbearing potential, pregnancy test is negative within 72 hours of first dose of study drug.
* if fertile, the patient agrees to use an effective method to avoid pregnancy for the duration of the study.
* Informed consent has been obtained.

Exclusion Criteria:

* No prior chemotherapy for metastatic or locally recurrent disease is allowed.
* Prio neo-adjuvant chemotherapy is allowed, and patients must have recovered from the acute toxicity of such therapies.

  * if a taxane was part of the adjuvant regimen, at least 12 months must have elapsed between the last dose of the taxane and the date of diagnosis of metastatic disease.
  * if a non-taxane-based adjuvant therapy was administered, at least six months must have elapsed between the last dose of the non- taxane-containing chemotherapy and the date of diagnosis of metastatic disease.
* Concurrent immunotherapy or hormonal therapy.
* Parenchymal brain metastases, including leptomeningeal involvement.
* Uncontrolled hypertension (defined as blood pressure of > 150/100 mmHg)
* NYHA Grade 2 or greater congestive heart failure
* History of coagulopathy, bleeding diathesis, therapeutic anticoagulation other than low dose or chronic ASA greater than or equal to 325 mg per day. Low dose coumadin for anticoagulation of venous access device or low dose molecular weight heparin (LMWH)for deep vein thrombosis prophylaxis or low dose (325 mg or less) ASA prophylaxis are allowed, but are best avoided if the treating physician feels it is safe to do so.
* Urine protein:creatinine ratio less than or equal to 1.0 at screening.
* No history of cerebrovascular accident within six months of study entry.
* Active symptomatic peripheral vascular disease (e.g. aortic aneurysm, claudication) within six months of study entry.
* Uncontrolled or severe cardiovascular disease including myocardial infarction or unstable angina within six months of study entry.
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal process within six months of study entry.
* No serious non-healing wound, ulcer, or bone fracture
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to first dose, or anticipation of need for major surgical procedure during the course of the study. No minor surgical procedure within seven days of study entry. Serious intercurrent medical or psychiatric illness, including serious active infection.
* History of other malignancy within the last 5 years which could affect the diagnosis or assessment of breast cancer.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Pregnant or nursing women.
* Patients with current sensory neuropathy of > Grade 1 will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2009-09-01 (Actual); Study Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Melbourne, Florida
  - Ocoee, Florida
  - Niles, Illinois
  - Terre Haute, Indiana
  - Columbia, Maryland
  - Westminister, Maryland
  - Saint Joseph, Missouri
  - Rochester, New York
  - Bedford, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Odessa, Texas
  - San Antonio, Texas
  - Tyler, Texas
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Salem, Virginia
  - Burien, Washington
  - Edmonds, Washington
  - Vancouver, Washington

REFERENCES:
- [Background] Danso M, et al. Phase II trial of weekly nab-paclitaxel in combination with bevacizumab as first-line treatment in metastatic breast cancer. Presented at 2008 ASCO Annual Meeting, May 30-June 3, 2008, Chicago, IL. Abstract No. 1075.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABI-007 Plus Bevacizumab
Started | 50
At Least One Response Assessment | 43
Completed | 24 (Treatment completed upon disease progression)
Not Completed | 26
Not completed — Unacceptable toxicity | 15
Not completed — Adverse Event | 4
Not completed — Physician Decision | 4
Not completed — Withdrawal by Subject | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | ABI-007 Plus Bevacizumab
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White, Non-Hispanic and Non-Latino | 40
  White, Hispanic or Latino | 7
  Other | 0
Weight [Mean (Standard Deviation); unit: kilograms] | 74.52 (15.430)
Menopausal status [Number; unit: participants]
  Pre-menopausal | 7
  Post-menopausal | 43
Eastern Cooperative Oncology Group (ECOG) status [Number; unit: participants] — ECOG status categories are defined as:
  * 0 (Fully Active)
  * 1 (Restrictive but Ambulatory)
  * 2 (Ambulatory but Unable to Work)
  * 3 (Limited Self-Care)
  * 4 (Completely Disabled)
  participants
    0 (Fully Active) | 23
    1 (Restrictive but Ambulatory) | 25
    2 (Ambulatory but Unable to Work) | 2
    3 (Limited Self-Care) | 0
    4 (Completely Disabled) | 0
Time from First Documented Metastasis/Relapse to Study Entry [Mean (Standard Deviation); unit: years] | 1.01 (3.123)
Dominant Current Site of Metastasis/Relapse [Number; unit: participants]
  Visceral | 49
  Non Visceral | 1

OUTCOME MEASURES:

1. Primary Outcome: Participants With At Least One Treatment-Emergent Adverse Event (TEAE)
Description: Count of study participants who had at least one treatment-emergent adverse event (TEAE) defined as any adverse event that began or worsened in grade after the start of study drug through 30 days after the last dose of study drug.
Time Frame: up to 25 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | ABI-007 Plus Bevacizumab
Number analyzed (Participants) | 50
participants | 50

2. Primary Outcome: Kaplan-Meier Estimates for Progression-free Survival
Description: Progression-free survival is defined as the time from first dose of study drug to the start of disease progression or patient death, whichever occurs first. Patients who do not have disease progression or have not died at the end of follow-up were censored at the last known time the patient was progression free. Patients that initiate other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
  Response Evaluation Criteria in Solid Tumors (RECIST) defines progressive disease (PD) as a >= 20% increase taking as reference the smallest sum of the longest diameters recorded since the treatment started; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: up to 39 months
Population: Treated population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007 Plus Bevacizumab
Number analyzed (Participants) | 50
months | 8.0 [5.3 to 10.3]

3. Secondary Outcome: Percentage of Participants With Objective Confirmed Complete or Partial Overall Response According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective response is complete response (CR) + partial response (PR). RECIST defines overall response of CR as the disappearance of all target and non-target lesions and no appearance of new lesions, confirmed at least 4 weeks after initial documentation. Overall response of PR is defined as >= 30% decrease from baseline in the sum of the longest diameters of target lesions and no progression of non-target lesions and no appearance of new lesions, confirmed at least 4 weeks after initial documentation. PR is also recorded when all measurable disease has completely disappeared, but a non-measurable component (i.e., ascites) is still present but not progressing and no appearance of new lesions. The objective response is determined by combining the response of target and non-target lesions and the appearance of new lesion(s) or not together.
Time Frame: up to 39 months
Population: Treated population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABI-007 Plus Bevacizumab
Number analyzed (Participants) | 50
percentage of participants
  Overall response (CR + PR) | 30 [17.3 to 42.7]
  Complete response (CR) | 0 [NA to NA] — not defined in analysis plan
  Partial response (PR) | 30 [NA to NA] — not defined in analysis plan

4. Secondary Outcome: Percentage of Participants With Stable Disease for >= 16 Weeks, or Complete or Partial Response According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Disease control is stable disease (SD) for >=16 weeks + complete response (CR) + partial response (PR). RECIST defines SD as neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease and no new lesions. Definitions for CR and PR can be found in outcome #3.
Time Frame: up to 39 months
Population: Treated population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ABI-007 Plus Bevacizumab
Number analyzed (Participants) | 50
percentage of participants
  CR + PR + SD>=16 weeks | 50 [36.1 to 63.9]
  Complete response (CR) | 0 [NA to NA] — not defined in analysis plan
  Partial response (PR) | 30 [NA to NA] — not defined in analysis plan
  Stable disease >=16 weeks (SD>=16 weeks) | 20 [NA to NA] — not defined in analysis plan

5. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response
Description: Duration of response is defined as progression-free survival in responders, i.e. as the time between the start of a complete response (CR) or partial response (PR) and the start of progressive disease (PD) or patient death from any cause, whichever occurred first. Patients that did not have progression or have not died were censored at the last known time the patient was progression free. Patients that initiate other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
  Progressive disease is defined in outcome #2. Complete response (CR) and partial response (PR) are defined in outcome #3.
Time Frame: up to 39 months
Population: Treated population of participants who had a response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007 Plus Bevacizumab
Number analyzed (Participants) | 15
months | 10.3 [9.0 to 20.8]

6. Secondary Outcome: Kaplan-Meier Estimates for Participant Survival
Description: Participant survival is the time from the first dose of study drug to patient death from any cause. Patients that did not die were censored at the last known time the patient was alive.
Time Frame: up to 39 months
Population: Treated population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ABI-007 Plus Bevacizumab
Number analyzed (Participants) | 50
months | 17.1 [13.7 to 23.8]

ADVERSE EVENTS:
Time Frame: up to 25 months
Arm/Group | ABI-007 Plus Bevacizumab
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 Plus Bevacizumab (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1 — Investigator evaluated the event as probably related to ABI.
Pneumonia (Infections and infestations) | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-007 Plus Bevacizumab (N=50)
Headache (Nervous system disorders) | 18
Neuropathy (Nervous system disorders) | 15
Neuropathy peripheral (Nervous system disorders) | 13
Peripheral sensory neuropathy (Nervous system disorders) | 13
Dizziness (Nervous system disorders) | 8
Dysgeusia (Nervous system disorders) | 8
Hypoaesthesia (Nervous system disorders) | 3
Paraesthesia (Nervous system disorders) | 3
Nausea (Gastrointestinal disorders) | 34
Diarrhoea (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 13
Abdominal distension (Gastrointestinal disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 31
Nail disorder (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 11
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 4
Nail discolouration (Skin and subcutaneous tissue disorders) | 4
Fatigue (General disorders) | 35
Oedema peripheral (General disorders) | 12
Asthenia (General disorders) | 9
Mucosal inflammation (General disorders) | 8
Pyrexia (General disorders) | 7
Pain (General disorders) | 6
Chills (General disorders) | 5
Infusion site pain (General disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 26
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 20
Anaemia (Blood and lymphatic system disorders) | 14
Leukopenia (Blood and lymphatic system disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Urinary tract infection (Infections and infestations) | 11
Upper respiratory tract infection (Infections and infestations) | 7
Cellulitis (Infections and infestations) | 3
Vulvovaginal mycotic infection (Infections and infestations) | 3
Hypertension (Vascular disorders) | 14
Hot flush (Vascular disorders) | 4
Hypotension (Vascular disorders) | 3
Lymphoedema (Vascular disorders) | 3
Insomnia (Psychiatric disorders) | 12
Anxiety (Psychiatric disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 9
Decreased appetite (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Vision blurred (Eye disorders) | 5
Conjunctivitis (Eye disorders) | 4
Lacrimation increased (Eye disorders) | 3
Dysuria (Renal and urinary disorders) | 6
Proteinuria (Renal and urinary disorders) | 4
Weight decreased (Investigations) | 4
Neutrophil count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Palpitations (Cardiac disorders) | 3

LIMITATIONS AND CAVEATS:
Interpretation of results is limited since the cell receptor subtype status of patients is not known.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it has been more than 2 years since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decided publication would hinder patent applications, Investigator must delay submission for up to 1 year. Investigator must delete confidential information before submission.